CLINICAL TRIAL: NCT02153385
Title: Effects of Yoga on Heart Rate Variability and Mood in Women: A Randomized Controlled Trial
Brief Title: Effects of Yoga on Heart Rate Variability and Mood in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, I-Hua Chu, PT, PhD, Assistant Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMU-Q099012
Record Dates: First submitted 2014-05-19; First posted 2014-06-03 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Heart Rate Variability
Keywords: Yoga, heart rate variability, stress, mood, women
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga group (Experimental): Two yoga sessions per week for 8 weeks
  Interventions: Other: Yoga
- Control group (No Intervention): Usual level of physical activity; no involvement in any yoga practice during the course of the study

INTERVENTIONS:
Other: Yoga — Yoga program was 60 min per session, twice per week for 8 weeks. Led by an experienced yoga instructor.
  Arms: Yoga group

SUMMARY:
Background: Women are more likely to suffer from depression and anxiety, which have been linked to reduced heart rate variability (HRV) and increased cardiovascular morbidity and mortality. The purpose of this study was to examine the effects of an 8-week yoga program on HRV and mood in generally healthy women. The investigators hypothesized that there would be improvements in HRV and reductions in perceived stress and symptoms of depression and anxiety after the yoga intervention.

Methods: Fifty-two healthy women were randomized to either a yoga group or a control group. Participants in the yoga group completed an 8-week yoga program, which comprised a 60-minute session, twice a week. Each session consisted of breathing exercises, yoga pose practice, and supine meditation/relaxation. Participants' HRV, perceived stress, depressive symptoms, and state and trait anxiety were assessed at baseline and week 9.

ELIGIBILITY:
Inclusion Criteria:

* women
* aged 18-50 years old
* body mass index < 30 kg/m2

Exclusion Criteria:

* currently engaged in regular yoga practice
* pregnant
* nursing
* had physical contraindications to exercise

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in heart rate variability at week 9 | The ourcome measure was assessed at baseline and at week 9
  Heart rate variability analysis was derived from continuous heart rate recording, at a sampling rate of 1024 Hz, using an electrocardiogram (ECG) system (MP 150, BIOPAC Systems, Goleta, CA, USA). Participants were instructed to avoid exercise one day before the assessment session and abstain from caffeinated food and beverages on the day of assessment. During the assessment, participants were instructed to relax in a supine position with no other tasks or stimulation for 20 minutes while the ECG was recording. The last 10 minutes of the ECG recording was analyzed for HRV. R-R intervals were computed and the HRV power spectrum was obtained via a fast Fourier transformation algorithm using an appropriate software program (HRV Analysis for Windows, version 1.1; Biosignal Imaging Group and Analysis, the University of Kuopio, Kuopio, Finland).

CONTACTS AND LOCATIONS:
Overall Officials: I-Hua Chu, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan